CLINICAL TRIAL: NCT05518903
Title: Quantitative In Vivo 68Ga-Fibroblast-Activation-Protein-Inhibitors (FAPI)-46 PET Imaging of Cancer-Associated Fibroblasts (CAFs) in Pancreatic Ductal Adenocarcinoma (PDA)
Brief Title: Investigational Scan (68Ga-FAPI-46 PET/CT) for Imaging of Cancer-Associated Fibroblasts for Localized Pancreatic Ductal Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MC220903; NCI-2022-06806 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-004884 (Other: Mayo Clinic Institutional Review Board); MC220903 (Other: Mayo Clinic); R01CA272628 (NIH)
Record Dates: First submitted 2022-08-24; First posted 2022-08-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Localized Pancreatic Adenocarcinoma; Resectable Pancreatic Ductal Adenocarcinoma; Stage 0 Pancreatic Cancer AJCC v8; Stage I Pancreatic Cancer AJCC v8; Stage IIA Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — FAPI-46; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (gallium GA 68 FAPi-46, PET/CT) (Experimental): Patients receive 68Ga-FAP-46 IV, then allow 60 minutes for 68Ga-FAPI-46 uptake. Patients then undergo PET/CT scans over 30 minutes at baseline (before SOC therapy), up to 2 scans approximately 8 weeks apart (at SOC re-staging visits), and a then a scan within 4 weeks of SOC surgical resection, if applicable.
  Interventions: Procedure: Computed Tomography; Drug: Gallium Ga 68 FAPi-46; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Gallium Ga 68 FAPi-46 — Given IV
  Other Names: 68Ga-FAPi-46; Gallium-68-FAPi-46
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial tests whether 68Ga-FAPI-46 positron emission tomography (PET)/computed tomography (CT) scan works to image cancer-associated fibroblasts (CAFs) in patients with pancreatic ductal adenocarcinoma (PDA) that has not spread to other parts of the body (localized). CAFs are a type of connective tissue cell that are found within or near cancerous tissue. Many CAFs express a protein called fibroblast activation protein (FAP) that are not found on healthy cells in large amounts. 68Ga-FAPI-46 is a radioactive chemical compound designed to circulate through the body and attach itself to FAP on PDA cells. A PET/CT scan is then used to detect the location of FAP lesions. PET scan is a procedure in which a small amount of radioactive glucose (sugar) is injected into a vein, and a scanner is used to make detailed, computerized pictures of areas inside the body where the glucose is taken up. Because cancer cells often take up more glucose than normal cells, the pictures can be used to find cancer cells in the body. CT scan is a procedure that uses a computer linked to an x-ray machine to make a series of detailed pictures of areas inside the body. The pictures are taken from different angles and are used to create 3-dimensional (3-D) views of tissues and organs. Combining a PET scan with a CT scan can help make the image easier to interpret. PET/CT scans are hybrid scanners that combine both modalities into a single scan during the same examination. Giving 68Ga-FAPI-46 PET/CT may help doctors improve upon the diagnosis and management of PDA.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the sensitivity and specificity of gallium Ga 68 FAPi-46 (68Ga-FAPI-46) PET for detection and quantification of cancer-associated fibroblasts (CAFs) in pancreatic ductal adenocarcinoma (PDA).

II. Construct, test and validate a model of surgical benefit or futility in potentially resectable PDA using 68Ga-FAPI-46 PET biomarkers in combination with other biomarkers of disease.

OUTLINE:

Patients receive 68Ga-FAP-46 intravenously (IV), then allow 60 minutes for 68Ga-FAPI-46 uptake. Patients then undergo PET/CT scans over 30 minutes at baseline (before standard of care [SOC] therapy), up to 2 scans approximately 8 weeks apart (at SOC re-staging visits), and a then a scan within 4 weeks of SOC surgical resection, if applicable.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years (yrs.) with treatment-naive biopsy-proven PDA or with findings diagnostic for PDA on baseline imaging (CT, MRI, or PET)
* Localized disease expected to undergo surgical resection following neoadjuvant therapy (NAT)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Ability to provide informed consent

Exclusion Criteria:

* Hypersensitivity to any excipients in 68Ga-FAPI-46
* Require emergency surgery
* Non-PDA histology on biopsy
* Histopathologically proven metastatic PDA
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of fibroblast-activation-protein-inhibitors (FAPI) positron emission tomography (PET) for detection and quantification of cancer-associated fibroblasts (CAFs) in pancreatic ductal adenocarcinoma (PDA) | Up to 5 years
  Using surgical immunohistochemistry (IHC) as gold standard.
Relationship between 68Ga-FAPI-46 PET metrics in PDA | Up to 5 years
  Relationship between 68Ga-FAPI-46 PET metrics assessed
Relationship between 68Ga-FAPI-46 PET metrics and cancer antigen 19-9 (CA19-9) biomarkers in PDA | Up to 5 years
  Relationship between 68Ga-FAPI-46 PET metrics and cancer antigen 19-9 (CA19-9) being assessed.
Relationship between 68Ga-FAPI-46 PET metrics and Kirsten rat sarcoma (KRAS), circulating tumor deoxyribonucleic acid (ctDNA) biomarkers in PDA | Up to 5 years
  Relationship between 68Ga-FAPI-46 PET metrics and Kirsten rat sarcoma (KRAS), circulating tumor deoxyribonucleic acid (ctDNA) being assessed.
Relationship between 68Ga-FAPI-46 PET metrics and staging examinations in PDA | Up to 5 years
  Relationship between 68Ga-FAPI-46 PET metrics and fludeoxyglucose F-18 (FDG) PET staging exam being assessed.
Relationship between 68Ga-FAPI-46 PET metrics and staging examinations in PDA | Up to 5 years
  Relationship between 68Ga-FAPI-46 PET metrics and magnetic resonance imaging (MRI) staging exam being assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ajit H. Goenka, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials